CLINICAL TRIAL: NCT01231815
Title: Coronary Flow Reserve Evaluation in PET and in MRI Scanner in Heart Transplanted Patients : Comparison With Multi-detectors Scanner
Acronym: RECOPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2008-007746-58
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Heart Disease
Keywords: Heart transplantation
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PET (Experimental): 15O-H2O PET
  Interventions: Radiation: 15O-H2O PET -
- MRI (Experimental): MRI
  Interventions: Radiation: MRI

INTERVENTIONS:
Radiation: 15O-H2O PET - — Assessment of coronary reserve using PET
  Arms: PET
Radiation: MRI — Assessment of coronary reserve using MRI
  Arms: MRI

SUMMARY:
Heart transplantation is the ultimate therapeutic option in patients with end-stage heart failure. Since advances in the treatment of acute rejection has increased early transplant survival, cardiac allograft vasculopathy (CAV) is the main factor limiting long-term survival. The prevalence of angiographically proven CAV is high, documented in 40-50% of transplant recipients 5 years after transplantation. Therefore, annual coronary angiography remains widely used to monitor transplanted patients, although pathologic studies and intravascular ultrasonography have demonstrated that coronary angiography underestimates the severity of CAV. Perfusion SPECT may underestimate allograft vasculopathy in case of diffuse coronary lesions. In this setting, the assessment of coronary reserve by means of Positron Emission Tomography (PET) and perfusion cardiac magnetic resonance imaging (CMR) have not been investigated.

DETAILED DESCRIPTION:
Aim of the study. The aim of the study is to compare the quantitative (using 15O-H2O PET) and semi-quantitative (using perfusion CMR) assessment of coronary reserve to the presence of coronary artery lesions documented by multidetector CT coronary angiography.

Methods. 30 patients with heart transplantation > 3 yrs will be included in two heart transplantation centers (Caen and Rouen university hospitals)

Expected results.

* To demonstrate that quantitative analysis of coronary reserve using 15O-H2O PET allows the assessment of cardiac allograft vasculopathy
* To establish the feasibility of adenosine stress CMR in this population
* To show a relationship between coronary lesions demonstrated using MDCT and the extent of coronary reserve impairment assessed using cardiac functional imaging (PET and CMR).

ELIGIBILITY:
Inclusion Criteria:

* Patient with heart transplantation > 3 years
* Candidate to a routine coronary angiography
* Age > 18 years old
* signed informed consent

Exclusion Criteria:

* Pregnancy or breast feeding women
* Recent acute coronary syndrome (<4weeks)
* High Blood Pressure ((SBP >=180 mmHg or DBP >=110 mmHg)
* Significant ventricular or supraventricular arrythmia
* Atrioventricular 2nd or 3rd degree blocks, long QT syndrome
* Standard contraindications to MRI including pacemaker/defibrillator, metallic clips on brain aneurysms, metal fragment in the eye etc...
* Congestive heart failure
* Hemodynamic instability
* Intolerance or contraindication to adenosine (history of asthma or bronchoplastic disease).
* Severe and known pulmonary artery hypertension
* Severe hypotension < 90 mmHg
* Contraindication to contrast iodinated media (allergy, patients with chronic renal failure with creatinine clearance < 50 ml/min, multiple myeloma, hyperthyroidism,...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
To compare the coronary flow reserve by a quantitative method (PET ... | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alain Manrique, MD, Principal Investigator — GIP Cyceron - CHU de Caen
Locations (2):
- France (2):
  - CHU de Caen - GIP Cyceron, Caen
  - CHU de Rouen, Rouen